CLINICAL TRIAL: NCT03459716
Title: Novel Screening Strategy for Systemic Sclerosis-associated Pulmonary Hypertension Incorporating Endothelial Biomarkers
Brief Title: Endothelial Biomarkers of Systemic Sclerosis-associated Pulmonary Hypertension
Acronym: BOSS-PH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Scleroderma Foundation (Unknown); Tulane University Health Sciences Center (Other); University Medical Center-New Orleans (Unknown)
Responsible Party: Principal Investigator, Matthew Lammi, Associate Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: IRB 10033SM
Record Dates: First submitted 2018-03-01; First posted 2018-03-09 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Scleroderma; Pulmonary Hypertension
Keywords: Biomarkers; Endothelial microparticles
MeSH Terms: conditions — Scleroderma, Diffuse; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic sclerosis patients w/ PH: Pulmonary hypertension will be defined as a mean pulmonary artery pressure≥25mmHg on right heart catheterization
  Interventions: Other: No intervention
- Systemic sclerosis patients w/o PH: Pulmonary hypertension will be excluded based on all of the following echocardiogram features: estimated systolic pulmonary artery pressure<35mmHg and absence of right atrial or right ventricular (RV) enlargement and lack of qualitative RV dysfunction. If a subject has any of these echo features, they will be referred for right heart catheterization (RHC) and included in the appropriate group based on their RHC results.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Systemic sclerosis (SSc, AKA scleroderma) is an autoimmune condition characterized by endothelial damage and progressive fibrosis of the skin and internal organs. One of the leading causes of morbidity and mortality in patients with SSc is pulmonary hypertension (PH), which is estimated to occur in up to 31% of high risk SSc patients. Early detection of patients with SSc-PH may lead to improved outcomes and although there have been concerted efforts to accurately screen for SSc-PH, these patients continue to present with advanced disease and suffer from poor survival. Therefore, better methods to screen for patients with PH and, perhaps more importantly, to screen for those at risk for PH development are desperately needed. Since PH and SSc are disorders originating from the endothelium, biomarkers that reflect endothelial damage are very promising tools to identify early disease. Such potential biomarkers include endothelial microparticles, asymmetric dimethylarginine (ADMA), pentraxin-3, and soluble endoglin. No previous study has used a combination of these biomarkers to detect the presence of PH in patients with SSc, or studied the novel concept of exercise-induced changes in biomarker levels. The investigators will collect the above listed endothelial biomarkers before and after exercise, and combine these levels with exercise echocardiogram findings, and routine clinical information to derive a composite detection score for the early identification of systemic sclerosis-associated PH.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >18 years 2. Meet American College of Rheumatology criteria for SSc

Exclusion Criteria:

1. Chronic kidney disease (estimated creatinine clearance <50mL/min)
2. Uncontrolled hypertension (diastolic blood pressure>120mmHg)
3. Acute coronary syndrome within the past 6 months
4. Chronic obstructive pulmonary disease
5. Diabetes mellitus
6. Hemolytic anemia
7. Active tobacco abuse

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 26 patients with systemic sclerosis-associated pulmonary hypertension and 26 patients with systemic sclerosis but no diagnosis of current pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite pulmonary hypertension detection score | At baseline
  A score will be derived by incorporating biomarkers, exercise echo results, pulmonary function tests, autoantibody status, 6-minute walk results, etc. into a linear regression model

SECONDARY OUTCOMES:
Composite pulmonary hypertension detection score | At 12 months
  A score will be derived by incorporating biomarkers, exercise echo results, pulmonary function tests, autoantibody status, 6-minute walk results, etc. into a linear regression model

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Lammi, MD, MSCR, Principal Investigator — LSU Health Sciences Center
Locations (1):
- University Medical Center-New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided